CLINICAL TRIAL: NCT01893645
Title: Pronto-7: Accuracy of Non-invasive Hemoglobin Measurement in Parturients
Acronym: Pronto-7
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: H12-00755
Record Dates: First submitted 2012-10-03; First posted 2013-07-09 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Hemoglobin Levels in Blood
Keywords: Pronto-7; SpHb; Obstetric patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women admitted to the British Columbia Women's Hospital for vaginal or cesarean delivery will get their Hb values spot-checked using the Pronto-7 device.
  Interventions: Device: Pronto-7

INTERVENTIONS:
Device: Pronto-7 — A new point-of-care pulse co-oximeter that offers a non-invasive and quick spot-checking of Hb (SpHb).

SUMMARY:
The measurement of blood hemoglobin (Hb) concentration is a routine procedure in pregnant women. The assessment of Hb involves several steps, including a needle stick, blood collection, blood sample analysis in the laboratory, and waiting for the results.

Pronto-7 (manufactured by Masimo, CA, USA) is a new portable device that allows a quick bedside Hb spot check. A finger clip probe, similar to the standard oxygen finger clip probe, provides hemoglobin values in less than 60 seconds.

In this prospective observational study the investigators will assess the clinical accuracy of Pronto-7 derived Hb values compared to the gold standard laboratory Hb values in obstetric patients. We will be calculating the mean difference between Pronto-7 and laboratory Hb values. We plan to recruit 55 pregnant women admitted for vaginal or cesarean delivery at BC Women's Hospital.

DETAILED DESCRIPTION:
Serum hemoglobin (Hb) concentration is one of the most common laboratory tests measured when a pregnant woman (parturient) is admitted for a vaginal or cesarean delivery. The Hb concentration is normally measured from a venous blood sample in clinical laboratories using co-oximetry.

A new point-of-care pulse co-oximeter, the Pronto-7 (Masimo Corporation, Irvine, CA, USA), is a portable device that offers a non-invasive and quick spot-checking of Hb (SpHb). Measurement with the Pronto-7 takes about 60 seconds and does not require the transfer of blood samples to a laboratory. In addition to SpHb, the device provides a perfusion index (PI) value (a numeric estimation of the pulse strength at the measurement site), heart rate, oxygen saturation, and finger temperature. Potential advantages of the Pronto-7 include reduced staff work, decreased exposure to potential biohazards, and reduced pain and discomfort to the patient.

A similar technology is used in Radical-7 pulse co-oximeter (Masimo Corporation, Irvine, CA, USA) for non-invasive Hb measurement. Radical-7 has been evaluated in human volunteers undergoing hemodilution, in patients undergoing spine surgeries, major urological procedures, and in critically ill patients. However, the results regarding the accuracy of this technology are conflicting.

ELIGIBILITY:
Inclusion Criteria:

* Are 19 - 40 years old
* Understand written and oral English
* Are greater than 37 weeks gestational age
* Have a singleton pregnancy

Exclusion Criteria:

* Have a laboratory Hb less than 100 g/L
* Have abnormal Hb disorders
* Have hyperbilirubinemia
* Have a peripheral vascular disease (e.g. Reynaud's syndrome)
* Have long or acrylic nails

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women admitted to the British Columbia Women's Hospital for vaginal or cesarean delivery (either elective or emergency).
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (Hb) value | 15-20 minutes before venipuncture
  Difference between the pre-venipuncture SpHb values and the laboratory Hb values (SpHb-Lab Hb difference) measured from the same extremity of each subject

SECONDARY OUTCOMES:
Comparisons of SpHb values | 15-20 minutes before venipuncture and 15-20 minutes after venipuncture
  Comparison between right and left hand SpHb values measured immediately before venipuncture.
  Comparison between right and left hand SpHb values measured immediately after venipuncture.
  Comparison of SpHb values measured from the same extremity immediately before and after venipuncture.
  Comparison of the SpHb-lab Hb differences between subjects in labour for vaginal delivery and subjects undergoing elective cesarean delivery.

OTHER OUTCOMES:
Consistency of lab Hb results | 4 hours after venipuncture
  Comparison between the first and second reading on the laboratory Cooximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gunka, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Macknet MR, Allard M, Applegate RL 2nd, Rook J. The accuracy of noninvasive and continuous total hemoglobin measurement by pulse CO-Oximetry in human subjects undergoing hemodilution. Anesth Analg. 2010 Dec;111(6):1424-6. doi: 10.1213/ANE.0b013e3181fc74b9. Epub 2010 Nov 3. PMID 21048100
- [Background] Miller RD, Ward TA, Shiboski SC, Cohen NH. A comparison of three methods of hemoglobin monitoring in patients undergoing spine surgery. Anesth Analg. 2011 Apr;112(4):858-63. doi: 10.1213/ANE.0b013e31820eecd1. Epub 2011 Mar 8. PMID 21385985
- [Background] Berkow L, Rotolo S, Mirski E. Continuous noninvasive hemoglobin monitoring during complex spine surgery. Anesth Analg. 2011 Dec;113(6):1396-402. doi: 10.1213/ANE.0b013e318230b425. Epub 2011 Sep 29. PMID 21965372
- [Background] Lamhaut L, Apriotesei R, Combes X, Lejay M, Carli P, Vivien B. Comparison of the accuracy of noninvasive hemoglobin monitoring by spectrophotometry (SpHb) and HemoCue(R) with automated laboratory hemoglobin measurement. Anesthesiology. 2011 Sep;115(3):548-54. doi: 10.1097/ALN.0b013e3182270c22. PMID 21716091
- [Background] Causey MW, Miller S, Foster A, Beekley A, Zenger D, Martin M. Validation of noninvasive hemoglobin measurements using the Masimo Radical-7 SpHb Station. Am J Surg. 2011 May;201(5):592-8. doi: 10.1016/j.amjsurg.2011.01.020. PMID 21545905
- [Background] Butwick A, Hilton G, Carvalho B. Non-invasive haemoglobin measurement in patients undergoing elective Caesarean section. Br J Anaesth. 2012 Feb;108(2):271-7. doi: 10.1093/bja/aer373. Epub 2011 Nov 23. PMID 22116296
- [Background] Gayat E, Aulagnier J, Matthieu E, Boisson M, Fischler M. Non-invasive measurement of hemoglobin: assessment of two different point-of-care technologies. PLoS One. 2012;7(1):e30065. doi: 10.1371/journal.pone.0030065. Epub 2012 Jan 6. PMID 22238693
- [Background] Sun J, Chernick MR, LaBudde RA. A bootstrap test for comparing two variances: simulation of size and power in small samples. J Biopharm Stat. 2011 Nov;21(6):1079-93. doi: 10.1080/10543406.2011.611082. PMID 22023677
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- See also: Related Info about the Pronto-7 Device — http://www.masimo.com/pronto-7/index.htm